CLINICAL TRIAL: NCT00048815
Title: Pharmacotherapy for Minor Depression
Brief Title: Drug Therapy to Treat Minor Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH); Office of Dietary Supplements (ODS) (NIH)
Responsible Party: Principal Investigator, Andrew A. Nierenberg, MD, Director Bipolar Clinic and Research Program, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01MH061758 (NIH); R01MH061758 (NIH); R01MH061757 (NIH); R01MH061394 (NIH); DSIR AT-SO; NCT00043524 (obsolete NCT alias); NCT00050544 (obsolete NCT alias)
Record Dates: First submitted 2002-11-08; First posted 2002-11-13 (Estimated); Results first posted 2018-05-11 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Depression
Keywords: Minor Depression; St. John's Wart
MeSH Terms: conditions — Depression | interventions — Citalopram; Dexetimide; Hypericum extract LI 160

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- citalopram (Active Comparator): Subjects in this arm received 20mg/day of citalopram taken orally for 12 weeks.
  Interventions: Drug: Citalopram
- St. John's Wort (Experimental): Subjects in this arm received 810 mg/day of St. John's Wort taken orally (in three tablets of 270mg each) for 12 weeks.
  Interventions: Drug: St. John's Wort
- Placebo (Placebo Comparator): Subjects in this arm received double-dummy (look-alike) placebo for 12 weeks.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Citalopram — Established Selective Serotonin Reuptake Inhibitor antidepressant
  Other Names: Celexa, Cipramil
  Arms: citalopram
Drug: St. John's Wort — Natural extract from the St. John's Wort plant.
  Other Names: Hypericum
  Arms: St. John's Wort
Drug: Placebos — Placebo pill
  Arms: Placebo

SUMMARY:
This 6-month study will compare the effectiveness of citalopram (Celexa®), hypericum (St. John's Wort), and placebo for the treatment of minor depression.

DETAILED DESCRIPTION:
Minor depression is highly prevalent, causes substantial morbidity and disability, presents a serious risk factor for the development of major depressive disorder, yet is under recognized and under treated. Researchers have determined that patients with minor depression frequently seek treatment from general practitioners and are often treated with prescription antidepressants. There is a need to evaluate the effectiveness of St. John's Wort in the management of minor depression. If the proposed study demonstrates the efficacy of St. John's Wort and/or citalopram, it will suggest treatment paradigms that can be tested and applied in primary care settings.

Subjects participated in a 12-week double-blind randomized study comparing St. John's Wort, citalopram, and placebo. Subjects were recruited through clinical referrals and community advertising. Data were obtained at the baseline visit (just prior to randomization) and at postrandomization visits conducted at 2-week intervals for the next 12 weeks, for a modified intent-to-treat sample consisting of all 73 subjects with at least 1 post-randomization visit (evaluable sample).

ELIGIBILITY:
Inclusion Criteria:

* Minor Depression symptoms for at least 6 months
* Endorse one of the DSM-IV "A" criteria for MDD and at least one other symptom of MDD or endorse both of the "A" criteria for MDD
* Global Assessment of Functioning (GAF) score < 70
* Short form health survey (SF-36) social functioning score <= 75% or an emotional role functioning score <= 67%
* HAM-D-17 score 10-17, inclusive
* Minor depression symptoms for at least 6 months

Exclusion Criteria:

* Major depressive disorder (MDD) or dysthymia within the past year or in partial remission of MDD
* At least a 12-week course of either citalopram at a minimum or 40 mg/day or St. John's Wort at a minimum of 900 mg/day during the current episode of depression
* Previous intolerance to either citalopram or St. John's Wort or history of nonresponse to either citalopram at a minimum of 40 mg/day or St. John's Wort at a minimum of 900 mg/day for at least 12 weeks
* Unstable medical illness, including cardiovascular, hepatic, renal, respiratory, endocrine, neurologic, or hematologic disease
* Uncontrolled seizure disorder
* The following DSM-IV diagnoses: organic mental disorders; substance use disorders, including alcohol, active within the last year or patients with a positive urine drug screen; schizophrenia; delusional disorder; psychotic disorders not elsewhere classified; bipolar disorder; bereavement; adjustment disorder; antisocial personality disorder; panic disorder, social phobia, generalized anxiety disorder (GAD), or obsessive compulsive disorder (OCD). Patients may have a lifetime diagnosis of an anxiety disorder as long as it is not current.
* Mood-congruent or mood-incongruent psychotic features
* Psychotropic drugs
* Hypothyroidism
* Investigational psychotropic drugs within the last year
* Positive toxicology screen
* Medications metabolized by the CYP3A4 system, where induction of this system poses a risk to the medical stability of the patient
* Pregnancy or refusal to use a medically accepted method of contraception
* Serious suicide or homicide risk
* Psychotherapy beginning less than 3 months ago

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2003-02; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew A. Nierenberg, M.D., Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Pittsburgh, Western Psychiatric Institute and Clinic, Pittsburgh, Pennsylvania

REFERENCES:
- See also: Click here to view the "Treatment for Minor Depression" NIH news release. — http://www.nimh.nih.gov/science-news/2003/treatment-for-minor-depression.shtml

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Citalopram | St. John's Wort | Placebo
Started | 24 | 26 | 23
Completed | 18 | 22 | 19
Not Completed | 6 | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Citalopram | St. John's Wort | Placebo | Total
Number analyzed (Participants) | 24 | 26 | 23 | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.3 (12.5) | 42.2 (14.1) | 51.4 (16.6) | 48.1 (15.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 11 | 37
  Male | 11 | 13 | 12 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 1 | 3
  Not Hispanic or Latino | 22 | 26 | 22 | 70
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 26 | 23 | 73

OUTCOME MEASURES:

1. Primary Outcome: Efficacy Assessed Using the Inventory of Depressive Symptomatology - Clinician Rated (IDS-C)
Description: We expect that subjects with minor depression treated for 12 weeks with St. John's Wort or citalopram will have significantly greater reduction in depressive symptom severity than those treated with placebo. This will be measured by blind ratings on the Inventory of Depressive Symptomatology - Clinician Rated (IDS-C) which has a total score range from 0 to 84 with 0 being not depressed at all and 84 being the most depressed. The change will be calculated by subtracting the Week 12 score from the Baseline score.
Time Frame: Change from Baseline to Week 12
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Citalopram | St. John's Wort | Placebo
Number analyzed (Participants) | 24 | 26 | 23
units on a scale | -11.47 (1.36) | -9.35 (1.23) | -10.49 (1.37)

2. Primary Outcome: Number of Adverse Events (Physical Symptoms) Emerging or Worsening During 12 Weeks of Treatment
Description: We expect that subjects treated for Minor Depression for 12 weeks with either St. John's Wort or citalopram will have similar safety profiles to subjects treated with placebo, and will not differ by more than 20% in rates of adverse side effects (e.g., nausea, headache, insomnia, hypersomnia, diarrhea) from subjects treated with placebo. This was measured by the number of adverse events (physical symptoms) emerging or worsening during 12 weeks of treatment.
Time Frame: Change from Baseline to Week 12
Measure: Mean (Standard Deviation); unit: Number of events
Arm/Group | Citalopram | St. John's Wort | Placebo
Number analyzed (Participants) | 24 | 26 | 23
Number of events | 4.7 (4.4) | 5.0 (4.5) | 3.4 (3.0)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: The Patient-Rated Inventory of Side Effects (PRISE; Rush et al., 2004) was administered at baseline and all subsequent visits. This obtained information not only about the presence or absence of 32 specific adverse events (and the opportunity to write in "others"), but whether those were present at a tolerable or distressing level or constituted a serious adverse event. Vital signs and medication compliance were also assessed at each visit during treatment.
Arm/Group | Citalopram | St. John's Wort | Placebo
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/26 | 0/23
Other Adverse Events (participants affected / at risk) | 23/24 | 22/26 | 18/23
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Citalopram (N=24) | St. John's Wort (N=26) | Placebo (N=23)
Diarrhea (Gastrointestinal disorders) | 8 (8) | 8 (8) | 1 (1)
Constipation (Gastrointestinal disorders) | 6 (6) | 8 (8) | 3 (3)
Dry Mouth (Gastrointestinal disorders) | 6 (6) | 6 (6) | 0 (0)
Nausea/Vomiting (Gastrointestinal disorders) | 6 (6) | 7 (7) | 4 (4)
Palpitations (Cardiac disorders) | 3 (3) | 3 (3) | 4 (4)
Dizziness on standing (Cardiac disorders) | 5 (5) | 4 (4) | 3 (3)
Chest Pain (Cardiac disorders) | 1 (1) | 1 (1) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 1 (1)
Increased perspiration (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1) | 1 (1)
Itching (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 10 (10) | 6 (6) | 11 (11)
Tremors (Nervous system disorders) | 4 (4) | 4 (4) | 0 (0)
Poor coordination (Nervous system disorders) | 1 (1) | 3 (3) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3) | 4 (4) | 5 (5)
Blurred vision (Eye disorders) | 5 (5) | 6 (6) | 4 (4)
Ringing in ears (Ear and labyrinth disorders) | 3 (3) | 1 (1) | 0 (0)
Frequent urination (Renal and urinary disorders) | 2 (2) | 3 (3) | 1 (1)
Menstrual irregularity (females) (Renal and urinary disorders) | 2/13 (2) | 0/13 (0) | 3/11 (3)
Difficulty sleeping (Nervous system disorders) | 10 (10) | 13 (13) | 7 (7)
Sleeping too much (Nervous system disorders) | 7 (7) | 5 (5) | 1 (1)
Loss of sexual desire (Reproductive system and breast disorders) | 7 (7) | 4 (4) | 5 (5)
Trouble achieving orgasm (Reproductive system and breast disorders) | 8 (8) | 5 (5) | 5 (5)
Trouble with erections (male) (Reproductive system and breast disorders) | 5/11 (5) | 1/13 (1) | 2/12 (2)
Anxiety (Psychiatric disorders) | 5 (5) | 5 (5) | 9 (9)
Poor concentration (Psychiatric disorders) | 6 (6) | 7 (7) | 7 (7)
General malaise (Psychiatric disorders) | 7 (7) | 2 (2) | 5 (5)
Restlessness (Psychiatric disorders) | 3 (3) | 8 (8) | 6 (6)
Fatigue (Psychiatric disorders) | 10 (10) | 3 (3) | 5 (5)
Decreased energy (Psychiatric disorders) | 9 (9) | 5 (5) | 5 (5)

LIMITATIONS AND CAVEATS:
Stringent inclusion criteria may have yielded a sample who depression was too mild to show added benefit for either active treatment beyond general therapeutic effects of study participation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No